CLINICAL TRIAL: NCT05317091
Title: The Effect of Laughter Yoga on Nurses' Perceived Stress Burnout and Life Satisfaction During the Pandemic Period: A Randomized Controlled Trial
Brief Title: The Effect of Laughter Yoga on Nurses' Perceived Stress Burnout and Life Satisfaction During the Pandemic Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Tülay KILINÇ, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: tulay24
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Abdominal Surgery; Hypertension; Done Laughter Yoga Before; Epilepsy
Keywords: Pandemic, Nurse, Stress, Burnout, Life satisfaction, Laughter yoga
MeSH Terms: conditions — Hypertension; Epilepsy; Burnout, Psychological; Personal Satisfaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Laughter yoga practice (Experimental): Laughter yoga for nurses The experimental group was divided into three groups as 18-17-16 people. Sessions 1st group Monday-Thursday between 12:00-13:00; 2nd group Tuesday-Friday between 17:00-18:00; The third group was held on Wednesday Saturday between 20:00-21:00.laughter yoga for nurses-Deep breathing exercises Deep breathing exercises (5 minutes), Warm-up exercises (10 minutes) laughter yoga for nurses-Childish games Childish games (10 minutes), Laughter exercises (15 minutes).
  Interventions: Other: Laughter yoga practiced
- Laughter yoga session parts-1 (Experimental): Deep breathing exercises (5 minutes) Breathing is held for 4-5 seconds after deep inspiration. While the arms are brought to the normal position, exhale slowly and rhythmically. When expressing after deep inspiration, the lips can be pursed as if whistling or exhaled with laughter.
  Interventions: Other: Laughter yoga practiced
- Laughter yoga session parts-2 (Experimental): Warm-up exercises (10 minutes) Rhythm of 1-2, 1-2-3 is added to increase the energy level even more and synchronize the movements of the group. After a few rhythmic clapping movements, another movement is added. Whisking hands left and right. Then an audible rhythm of ho, ho, ha-ha-ha is added to the clapping gesture. Make eye contact with people in the group and smile at them.
  Interventions: Other: Laughter yoga practiced
- Laughter yoga session parts-3 (Experimental): Childish games (10 minutes) Childlike games are used to help laugh without reason just like a child. The group is motivated by visualizing these games in their minds, raising the arms up in the form of a "Y" letter, and saying "very good (applause), very good (applause), hey" with palms facing the sky.
  Interventions: Other: Laughter yoga practiced
- Laughter yoga session parts-4 (Experimental): Laughter exercises (15 minutes) This section includes a variety of laughter exercises such as greetings, strawberry milk, conductor, bonus, hot soup, lion, aloha, bird, appreciation, laughter lotion, elevator, cream cake, and bursting balloon laughter.
  Interventions: Other: Laughter yoga practiced

INTERVENTIONS:
Other: Laughter yoga practiced — In this study, 8 sessions of laughter yoga were applied to the nurses in the experimental group as an intervention, twice a week for 4 weeks. Due to the Covid-19 pandemic; Laughter Yoga sessions were held on the web through the 'ZOOM' program.
  For this reason, it is recommended that the laughter yoga sessions be done with a group and that the group should consist of at least five people in order to provide group dynamics. Sessions are planned according to the days and hours that nurses can attend. Sessions 1st group Monday-Thursday between 12:00-13:00; 2nd group Tuesday-Friday between 17:00-18:00; The third group was held on Wednesday-Saturday between 20:00-21:00. The nurses were constantly contacted (whatsapp, phone) to ensure that they attend the sessions regularly and that there is no interruption in the sessions. No experiment was performed on the control group during the study. However, after the research, a 4-week laughter yoga was given to the nurses who wanted it.

SUMMARY:
This study aimed to determine the effects of laughter yoga on the perceived stress, burnout and life satisfaction of nurses working actively during the pandemic period. A total of 120 nurses, determined by power analysis, were included in the randomized controlled study. The study included 2 groups. (A group of nurses who have active contact with patients diagnosed with or at risk of covid-19, group B: nurses who have active contact with patients diagnosed with or at risk of covid-19 and participate in laughter yoga practice. Laughter yoga; immune system antibodies and endorphin hormone. It has been proven by experimental studies that there is a connection between the two, that it has a healing effect, that it accelerates the circulatory system as an adverse effect to stress, and that it has a vasodilation effect in the vessels.

DETAILED DESCRIPTION:
The study data were collected by the researchers using online systems with the snowball method due to the pandemic. The inclusion criteria of the study (not having undergone abdominal surgery in the last three months, not having uncontrolled hypertension, not having glaucoma, hernia, epilepsy, not having received a psychiatric diagnosis-treatment, not having received a diagnosis-treatment for sleep problems, having done laughter yoga before) The study consisted of 100 nurses who agreed to participate in the study. Introductory features form consisting of 13 questions, Maslach Burnout Scale and Life Satisfaction Scale, Perceived Stress Scale and life satisfaction scale were used to collect data. Research data were collected in 3 months. During the study, 9 people from the experimental group (8 people did not attend the sessions regularly, 1 person left voluntarily), 10 people from the control group (he left voluntarily) quit the study. Finally, the research was completed with 101 nurses, 51 of whom were in the experimental group and 50 in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Not have undergone abdominal surgery in the past three months
* Uncontrollable hypertension
* Without epilepsy

Exclusion Criteria:

* Antidepressant etc. nurses using drugs
* Not attending sessions regularly

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form (questionnaire) | up to 2 weeks
  In this form prepared by the researchers; There are a total of 9 questions including age, gender, education level, marital status, working year, frequently worked shift, Covid-19 passing and being vaccinated, whether or not he has knowledge about laughter yoga.
Perceived Stress Scale | up to 5 weeks]
  The scale, which was created in order to understand how stressful individuals perceive certain events they experience, consists of 14 items, graded in a 5-point Likert type. In the scale, 7 items containing positive statements are reverse scored. The score range of the scale ranges from 0 to 56, and a high score indicates a high level of stress. The internal consistency coefficient of the scale was calculated as 0.84. In this study, the Cronbach alpha internal consistency coefficient was found to be 0.75.
Maslach Burnout Scale | up to 5 weeks
  The scale, consisting of 22 items and three sub-dimensions, is in the 5-point Likert type. The sub-dimensions of the scale are emotional exhaustion, depersonalization and personal achievement. Positive statements in the dimension of personal achievement are reverse coded. The high mean score of the emotional exhaustion and depersonalization sub-dimensions and low personal achievement mean scores indicate high burnout. The lowest score that can be obtained from the scale is 0 and the highest score is 88. The Cronhbach Alpha values of the scale were found to be 0.83 for emotional exhaustion, 0.65 for depersonalization and 0.72 for personal achievement.
Life Satisfaction Scale | up to 5 weeks
  There are 5 items in the scale, and each item is arranged according to a 7-point answer system. A score between 5-35 can be obtained from the scale. Higher scores indicate higher life satisfaction. The Cronbach Alpha value of the scale is .88. In this study, the Cronbach Alpha coefficient was found to be .87.

SECONDARY OUTCOMES:
Perceived Stress Scale | up to 5 weeks
  The scale, which was created in order to understand how stressful individuals perceive certain events they experience, consists of 14 items, graded in a 5-point Likert type. In the scale, 7 items containing positive statements are reverse scored. The score range of the scale ranges from 0 to 56, and a high score indicates a high level of stress. The internal consistency coefficient of the scale was calculated as 0.84. In this study, the Cronbach alpha internal consistency coefficient was found to be 0.75.
Maslach Burnout Scale | up to 5 weeks
  The scale, consisting of 22 items and three sub-dimensions, is in the 5-point Likert type. The sub-dimensions of the scale are emotional exhaustion, depersonalization and personal achievement. Positive statements in the dimension of personal achievement are reverse coded. The high mean score of the emotional exhaustion and depersonalization sub-dimensions and low personal achievement mean scores indicate high burnout. The lowest score that can be obtained from the scale is 0 and the highest score is 88. The Cronhbach Alpha values of the scale were found to be 0.83 for emotional exhaustion, 0.65 for depersonalization and 0.72 for personal achievement.
Life Satisfaction Scale | up to 5 weeks
  There are 5 items in the scale, and each item is arranged according to a 7-point answer system. A score between 5-35 can be obtained from the scale. Higher scores indicate higher life satisfaction. The Cronbach Alpha value of the scale is .88. In this study, the Cronbach Alpha coefficient was found to be .87.

CONTACTS AND LOCATIONS:
Locations (1):
- Tülay Kılınç, Erzurum, Palandöken, Turkey (Türkiye)

REFERENCES:
- [Derived] Si S Celi K A, Kilinc T. The effect of laughter yoga on perceived stress, burnout, and life satisfaction in nurses during the pandemic: A randomized controlled trial. Complement Ther Clin Pract. 2022 Nov;49:101637. doi: 10.1016/j.ctcp.2022.101637. Epub 2022 Jul 5. PMID 35810525